CLINICAL TRIAL: NCT06987175
Title: Effects of Sedante Neo Therapy on Pain, Range of Motion and Quality of Life in Patients With Non Specific Low Back Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0134
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain; Range of Motion; Pain
Keywords: sedante neo therapy; non specific low back pain; quality of life
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional exercises (Experimental): receive conventional exercises only. Conventional exercises will be performed for 20 minutes, each exercise will be performed 20 times with 10 seconds hold.
  Interventions: Other: Conventional exercises
- Sadante neo therapy (Experimental): SAN machine having 3 tube cords on both sides. Each tube cord contains 2 pairs of flat suction cups. We will use 4 pair of flat suction cups in this study. We will place 2 pair on left and two on right para spinal muscles of lumber in prone lying. Due to its automatic suctioning capability, these cups can easily stick to skin. After placing the cups on lumber each patient of group A will receive its stimulation for about 10 minutes every day for about 4 weeks along with conventional exercises.
  Interventions: Other: sadante neo therapy

INTERVENTIONS:
Other: sadante neo therapy — SAN machine having 3 tube cords on both sides. Each tube cord contains 2 pairs of flat suction cups. We will use 4 pair of flat suction cups in this study. We will place 2 pair on left and two on right para spinal muscles of lumber in prone lying. Due to its automatic suctioning capability, these cups can easily stick to skin. After placing the cups on lumber each patient of group A will receive its stimulation for about 10 minutes every day for about 4 weeks along with conventional exercises.
  Arms: Sadante neo therapy
Other: Conventional exercises — receive conventional exercises only. Conventional exercises will be performed for 20 minutes, each exercise will be performed 20 times with 10 seconds hold.
  Arms: conventional exercises

SUMMARY:
this study is to evaluate the effects of SADANTE neo therapy on pain, range of motion and quality of life in patients with non-specific low back pain.

DETAILED DESCRIPTION:
This study is to evaluate SADANTE neo therapy on pain, range of motion and quality of life in patients with low back pain. This study will identify the effects that will help the physiotherapists in making the treatment plan for low back pain. This can be an alternative non pharmacological therapy to improve the quality of pain management with maximum benefits and minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 20 yeras to 40 years.

  * Both male and female included.
  * Having non-specific low back pain.
  * Having SF-MPQ score 1and 2 (1 means mild, 2 means moderate)
  * Having ODI score 5 to 24
  * Having SF-36 healty survey score below 50
  * Having range of motion below normal.

Exclusion Criteria:

* Below 20 years and above 40 years patient are excluded
* Cervical, knee pain and other conditions excluded.
* Children are excluded
* Red flags ( tuberculosis, carcinoma heart disease etc) excluded

  -Open sores
* Psychiatric diseases such as depression, phobias

  * Patient with history of surgery in lumber region

Ages: 20 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire: | 4th week
  The McGill Pain Questionnaire can be used to evaluate a person experiencing significant pain. It can be used to monitor the pain over time and to determine the effectiveness of any intervention.

SECONDARY OUTCOMES:
Oswestry disability index: | 4th week
  This questionnaire has been designed to give us information as to how your back pain has affected your ability to manage everyday life
Rand 36-items helath survey | 4th week
  The rand 36-items survey is used to indicate the health status of particular populations, to help with service planning and to measure the impact of clinical and social interventions

CONTACTS AND LOCATIONS:
Overall Officials: Ameena Amjad, Phd, Principal Investigator — Riphah International University
Locations (1):
- Arthritis and pain care clinic Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ceballos-Laita L, Jimenez-Del-Barrio S, Marin-Zurdo J, Moreno-Calvo A, Marin-Bone J, Albarova-Corral MI, Estebanez-de-Miguel E. Comparison of dry needling and self-stretching in muscle extensibility, pain, stiffness, and physical function in hip osteoarthritis: A randomized controlled trial. Complement Ther Clin Pract. 2022 Nov;49:101667. doi: 10.1016/j.ctcp.2022.101667. Epub 2022 Sep 11. PMID 36152527
- [Background] Iglesias-Gonzalez JJ, Munoz-Garcia MT, Rodrigues-de-Souza DP, Alburquerque-Sendin F, Fernandez-de-Las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in patients with chronic nonspecific low back pain. Pain Med. 2013 Dec;14(12):1964-70. doi: 10.1111/pme.12224. Epub 2013 Aug 15. PMID 23947760
- [Background] Facci LM, Nowotny JP, Tormem F, Trevisani VF. Effects of transcutaneous electrical nerve stimulation (TENS) and interferential currents (IFC) in patients with nonspecific chronic low back pain: randomized clinical trial. Sao Paulo Med J. 2011;129(4):206-16. doi: 10.1590/s1516-31802011000400003. PMID 21971895